CLINICAL TRIAL: NCT05868005
Title: Delivering an Innovative Multi-disease Screening Tool to High-risk Migrant Populations
Brief Title: Delivering a Multi-disease Screening Tool to Migrant Populations
Acronym: ISMiHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barcelona Institute for Global Health (Other)
Collaborators: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Distrito Sanitario Poniente de Almería (Unknown); Hospital de Poniente (Unknown); Universidad de Granada (Other); Consorci d'Atenció Primària de Salut de l'Eixample (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PI21/00651
Record Dates: First submitted 2023-04-17; First posted 2023-05-22 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2024-09

CONDITIONS: Hiv; Hepatitis B; Hepatitis C; Tuberculosis; Chagas Disease; Schistosomiasis; Strongyloidiasis; Female Genital Mutilation Type I Status; Female Genital Mutilation Type II Status; Female Genital Mutilation Type III Status
Keywords: Screening; Migrant; Clinical decision support system; Digital software tool; Electronic patient record system; Primary care; Individual risk assessment; HIV; Hepatitis B; Hepatitis C; Tuberculosis; Chagas Disease; Schistosomiasis; Strongyloidiasis; Female genital mutilation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis B; Hepatitis C; Tuberculosis; Chagas Disease; Schistosomiasis; Strongyloidiasis | interventions — Primary Health Care

STUDY DESIGN:
Intervention Model Description: A pragmatic cluster controlled randomised trial will be conducted in 35 PCCs in Catalonia. The randomization will be performed through a statistical software for each pair of selected health centres, stratified by study area and by density of migrant population in the area (low, medium and high). For each pair of PCCs, one PCC will be randomly selected to implement the screening program through the ISMiHealth software, and it will be compared with the other PCC, which will follow the current routine care practices. In both cases, health professionals will receive a training session on migrant health; the contents will include, for each condition, epidemiological aspects, diagnosis, treatment, and the screening recommendation. Around 980 health professionals will participate as software users but the exact number may vary due to replacements, sick leaves, rotations, etc. In Andalusia, a pilot cluster randomized trial will be carried out to evaluate preliminary effectiveness data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary care centres with the ISMiHealth software tool. (Experimental): Primary care centres implementing the screening programme through the ISMiHealth software (tool-based arm).
  Interventions: Other: Clinical decision support system for screening of migrants using the ISMiHealth software tool.
- Primary care centres that follow current routine care. (No Intervention): Primary care centres that follow the current practices in routine care (non tool-based arm).

INTERVENTIONS:
Other: Clinical decision support system for screening of migrants using the ISMiHealth software tool. — The implementation of the screening programme will be facilitated using a simple and user-friendly software tool (ISMiHealth).
  When an individual attends the PCC for any reason, the tool will generate an alert for health professionals in the EPR system, with recommendations on the conditions that should be considered for screening, based on this patient's characteristics (country of birth, age and sex). Health professionals will decide what diseases/conditions should be screened for, supported by the recommendations of the digital software (intervention centres) or based on their knowledge on the epidemiological background of the diseases (control centres). In any case, health professionals will be responsible for requesting serology tests, chest radiographies and/or referrals to specialists.
  Other Names: Former intervention: Screening migrant patients using a computer tool adapted to clinical histories in primary care (CRIBMI).; Former acronym of current study: INNoMiGs
  Arms: Primary care centres with the ISMiHealth software tool.

SUMMARY:
Migrants' overall health status may be improved by increasing the detection of certain infectious diseases and other conditions for which effective care is available. This can be achieved through a systematic screening of these conditions using innovative and digital solutions implemented in routine health care.

This study aims to evaluate the implementation of a screening programme for migrants at primary care level in two different settings of Spain (Catalonia and Andalusia) using an innovative digital and user-friendly software tool (ISMiHealth). In Catalonia, the ISMiHealth tool has already been integrated into the Electronic Patient Record (EPR) system (eCAP) as part of a pilot study in 2018; currently, the research team aims to validate the tool in a higher number of primary care centres in this area. Therefore, a pragmatic cluster randomised controlled trial will be conducted with two parallel groups, in which selected centres using the novel software ISMiHealth will be compared to others that follow the current routine practice. On the other hand, in Andalusia a pilot cluster randomised controlled trial will be carried out, where the ISMiHealth tool will be implemented in the EPR system (DIRAYA) to evaluate the preliminary effectiveness of the tool in other settings.

The ISMiHealth software is a clinical decision support system that provides recommendations for primary healthcare professionals on screening for targeted conditions. It currently includes: 7 communicable diseases (Human immunodeficiency virus, Hepatitis B and C virus, Tuberculosis, Chagas diseases, strongyloidiasis and schistosomiasis) and one key health condition (female genital mutilation). Through routinely collected variables (country of birth, age, and sex), the software performs an individualised risk assessment and provides real-time prompts to healthcare professionals on screening for the selected health conditions. In any case, health professionals will be responsible for requesting screening tests and/or referrals to specialists.

DETAILED DESCRIPTION:
1. Objectives

   General objective: To develop an integrated and primary care based, communicable diseases and female genital mutilation (FGM) screening programme for migrant populations in Spain in order to promote better health and integration.

   Specific objectives:
   * Aim 1: To develop a Spanish consensus guidance on migrant screening recommendations based on existing European examination/screening programmes and on a consensus of a country-expert transdisciplinary national collaborative network.
   * Aim 2: To scale-up and validate a simple and user-friendly innovative digital tool that will be integrated into the local electronic patient record (EPR) system of primary care in two different settings (Catalonia and Andalusia), and that aims to facilitate targeted screening to migrants presenting for a routine appointment. This digital tool will support health professionals to follow best-practice recommendations, while considering patients' individual characteristics (country of birth, age, sex) and therefore specific risk factors.
2. Study design

   This study will be developed into two sub-studies in order to accomplish the specific objectives.

   2.1 Study 1 related to aim 1. Spanish consensus guidance on migrant screening recommendations.
   1. A comparative review and analysis of existing screening programmes at regional, national and international level will be performed.
   2. A report with the reviewed results will be developed and presented in the consensus workshops.
   3. A consensus workshop with national experts will be carried out by study site to establish which diseases will be included in the final screening algorithm and what will be defined as the screening criteria for each condition. The tentative elements to include are Human immunodeficiency virus (HIV), Hepatitis B virus (HBV), Hepatitis C virus (HCV), Tuberculosis (TB), selected parasitic infections and FGM. For most of the communicable diseases, the screening criteria will be fully aligned with the current European Centre for Disease Prevention and Control (ECDC) screening guidelines and recommendations.
   4. To measure the level of agreement with the recommendations, a questionnaire based on a Likert Scale of 5 points (1- Strongly disagree, 2- Disagree, 3- Neutral, 4- Agree and 5- Strongly agree) will be sent to the different experts invited to the workshops.

   2.2 Study 2 related to aim 2. Operational implementation of a screening programme using the ISMiHealth software and evaluation of its impact and equity.
   1. Study design and subjects. A pragmatic cluster randomised controlled trial will be conducted in 35 Primary care centers (PCCs) of Catalonia to explore and assess the effectiveness of the software tool ISMiHealth [see sample size calculation in the Statistical Analysis Plan (SAP)]. The screening programme will be implemented in a real-life context in the selected PCCs, and the receivers/users of the tool will be all health professionals (general practitioners and nurses) working at the intervention centres. On the other hand, the tool and the outcomes of the study will be evaluated in the migrant patients, the indirect beneficiaries of the tool. Additionally, a pilot clustered randomised controlled trial will be conducted in Andalusia, implementing the screening programme in six PCCs to explore preliminary effectiveness data.

      In the site of Catalonia approximately 840 health professionals will participate in the intervention while in Andalusia approximately 140 health professionals will participate.

      ISMiHealth set a series of rules that provide real-time prompts to health professionals on screening of infectious diseases and FGM in migrants. Therefore, when an individual comes to the PCC for any reason, the health professional will receive a message in the EPR system, inserted as a pending task assignment, with a recommendation on the conditions that should be considered for screening. For this, the software will perform an individual risk-assessment based on the patient's background characteristics (country of birth, age and sex). The software tool is also able to identify if a person had already a diagnosis of any of the conditions included in the algorithm [based on the International Classification Diagnosis codes, Ninth version (ICD-9) or Tenth version (ICD-10)] or if a diagnostic test had been performed for any condition included in the program. In such cases, the automated electronic prompt does not appear for that condition.

      Before the intervention, we will hold training sessions with the same screening recommendations for both the intervention and control centres but the latter ones will not initiate the tool/prompts onto the EPR system. In addition, a pilot test will be conducted with 3 health professionals to assure the correct functioning of the tool. At last, the ISMiHealth software will be implemented in the EPR systems of the participating PCCs.
   2. Implementation strategy. During the implementation phase, real-time monitoring of the strategy will be performed (by a data manager and a study coordinator from each PCC) in order to identify opportunities for improvement and optimization of the process. The technical monitoring will help identify errors in the implementation of the alerts in the EPR system, to be mitigated in real-time. Quantitative indicators will also be provided by the Information Service of the Primary Care Services (SISAP) to evaluate the outcomes of the implementation.
3. Intervention

   The implementation of the screening programme will be facilitated using a simple and user-friendly tool that helps health professionals to follow best-practice recommendations while taking into account patients' individual characteristics: country of birth , age, sex.

   In Catalonia, the digital tool has already been integrated into the EPR system (eCAP), a program shared by all PCCs that are part of the Catalan Institute of Health, as part of a pilot study. The three demographic variables (country of birth, age, and sex) are routinely collected by the PCCs' administrative staff and documented in electronic medical records. Once the administrator collects these variables in the computer system, the tool will generate an alert that will be reflected once the patient's medical history is reopened.

   In Andalusia, the software tool will be generated from demographic data stored in the Database of Users of the Andalusian Health Service (SAS, as its Spanish acronym). Once the health professional accesses the digital tool, he/she will have to mark in a check-list produced by the tool the conditions that the patient has already been screened for. In both study sites, the data of the patients is not registered nor collected by the tool, it is only used to produce the alert.
4. Data analysis

Since the ISMiHealth tool is in different phases of implementation in each site, and the algorithms are based on different recommendations, there will be two independent data analyses: i) in Catalonia, the health impact of the tool will be evaluated in 35 PCCs; and ii) in Andalusia, the preliminary effectiveness data will be estimated in the six PCCs where the tool will be pilot tested. See SAP attached.

ELIGIBILITY:
I) PCCs

Inclusion criteria:

• Centres with a migration density higher than 7%.

II) Primary care professionals

Inclusion criteria:

• Aged >18 years old working at the selected PCCs.

III) Migrant populations

Inclusion criteria:

* Individuals assigned to a PCC.
* Patients attending the PCCs for any reason.
* Aged >15 years old in the Catalonian site.
* Aged >14 years old in the Andalusian site.
* Coming from countries in the geographic areas of Africa, Latin-America, Asia and Eastern Europe following the categorization of the United Nations Statistical Commission.

Exclusion criteria:

* For the active TB recommendation, migrants residing in the host country for more than five years.
* For FGM recommendation, being a male.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 980 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the detection rate per month of all aggregated infections (HIV, HBV, HCV, TB, T.cruzi, S.stercoralis and Schistosoma spp. infections) between the intervention and control centres | Over at least 5 years until the end of the intervention (1 year).
  In the Andalusian site, syphilis, latent TB and intestinal parasites will also be included. The monthly detection rate will be based on positive serologies, chest radiographies, the ICD-9 (for Andalusia) or ICD-10 (for Catalonia) of FGM and/or gynaecologist referrals, within the migrant patients who visited their assigned centre during the intervention period. Also, positive tuberculin skin test (TST) and/or Interferon Gamma Release Assay (IGRA) and stool samples will be considered for the Andalusian site. Control and intervention PCCs will be compared before and after the implementation.

SECONDARY OUTCOMES:
Comparison of the detection rate per month of each individual condition, the infections and FGM cases, between the intervention and control centres | Over at least 5 years until the end of the intervention (1 year).
  The monthly detection rate will be based on positive serologies, chest radiographies, ICD-9/ICD-10 of FGM and/or gynaecologist referrals, TST/IGRA and stool samples (for Andalusia), within the migrant patients who visited their assigned centre during the intervention period. Control and intervention PCCs will be compared before and after the implementation.
Comparison of the number of early HIV diagnoses | Over at least 5 years until the end of the intervention (1 year).
  The number of early diagnoses of HIV will be assessed using the CD4 cell count of migrant patients diagnosed with an HIV infection. The early diagnoses will be compared between the control and intervention PCCs before and after the implementation. If possible, we will estimate the monthly detection rate of early diagnoses and also compare it between the intervention and control PCCs.
Comparison of the number of early HBV and HCV diagnoses | Over at least 5 years until the end of the intervention (1 year).
  The number of early diagnoses of HBV and HCV will be assessed using the levels of transaminases, platelets, bilirubin, and clotting parameters from blood analyses of migrant patients diagnosed with HBV or HCV. The early diagnoses will be compared between the control and intervention PCCs before and after the implementation. If possible, we will estimate the monthly detection rate of early diagnoses and also compare it between the intervention and control PCCs.
Comparison of the number of screening tests performed for all aggregated infections | Over at least 5 years until the end of the intervention (1 year).
  The number of the screening tests performed for all aggregated infections (serological tests, chest radiographies, TST or IGRA tests and stool samples in the case of the Andalusian site) will be compared between the intervention and control PCCs before and after the implementation.
Comparison of the the number of screening tests performed for each individual condition | Over at least 5 years until the end of the intervention (1 year).
  The number of the screening tests performed for each individual condition will be compared between the intervention and control PCCs before and after the implementation.
Associations between the screening performance of all aggregated infections (yes/no) and patients' age (in years) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of the aggregated infections (yes-if the patient has been tested for at least one of the seven infections during the study period/no-if the patient was not tested) as the outcome variable and patients' age as the predictor variable.
Associations between the screening performance of all aggregated infections (yes/no) and the time that patients have been registered in the Spanish National Health System (in years) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of the aggregated infections (yes-if the patient has been tested for at least one of the seven infections during the study period/no-if the patient was not tested) as the outcome variable and time registered in the Spanish Health System as the predictor variable.
Associations between the screening performance of all aggregated infections (yes/no) and patients' sex (female/male) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of the aggregated infections (yes-if the patient has been tested for at least one of the seven infections during the study period/no-if the patient was not tested) as the outcome variable and patients' sex as the predictor variable.
Associations between the screening performance of all aggregated infections (yes/no) and patients' area of birth (Africa/Latin America/Asia/Eastern Europe) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of the aggregated infections (yes-if the patient has been tested for at least one of the seven infections during the study period/no-if the patient was not tested) as the outcome variable and patients' area of birth as the predictor variable. The areas of birth will be based in the geographical division of the United Nations Statistical Division.
Associations between the screening performance of all aggregated infections (yes/no) and the region where the PCC is located (Terres de l'Ebre/Lleida/Tarragona/Costa de Ponent) will be analysed using the data collected in the SISAP database | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of the aggregated infections (yes-if the patient has been tested for at least one of the seven infections during the study period/no-if the patient was not tested) as the outcome variable and the region of the PCC as the predictor variable.
Associations between the screening performance of all aggregated infections (yes/no) and the type of region where the PCC is located in Catalonia, Spain (urban/rural) will be analysed using the data collected in the SISAP database | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of the aggregated infections (yes-if the patient has been tested for at least one of the seven infections during the study period/no-if the patient was not tested) as the outcome variable and the type of region of the PCC as the predictor variable.
Associations between the screening performance of all aggregated infections (yes/no) and if the patient fulfilled the criteria of the screening recommendation (yes/no) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of the aggregated infections (yes-if the patient has been tested for at least one of the seven infections during the study period/no-if the patient was not tested) as the outcome variable and fulfilled the criteria of the screening recommendation (yes- if the patient had the criteria of being tested for at least one infection, criteria generated by the algorithm of the ISMiHealth software using the variables country of birth, age and sex/no- if the patient did not meet the criteria) as the predictor variable.
Associations between the screening performance of all aggregated infections (yes/no) and the arm of the study (Intervention/Control) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of the aggregated infections (yes-if the patient has been tested for at least one of the seven infections during the study period/no-if the patient was not tested) as the outcome variable and the arm of the study as the predictor variable.
Associations between the screening performance of all aggregated infections (yes/no) and patients' immunosuppression status (yes/no) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of the aggregated infections (yes-if the patient has been tested for at least one of the seven infections during the study period/no-if the patient was not tested) as the outcome variable and patients' immunosuppression status (yes- if the patient has an ICD-code diagnosis of an immunosuppressive disorder and/or have a prescription of an immunosuppressive drug/no- if the patient is not immunosuppressed) as the predictor variable.
Associations between the screening performance of all aggregated infections (yes/no) and the presence of another condition (yes/no) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of the aggregated infections (yes-if the patient has been tested for at least one of the seven infections during the study period/no-if the patient was not tested) as the outcome variable and the presence of another condition (yes- if the patient has an ICD-code of another condition [co-morbidity]/no- if the patient does not present another condition) as the predictor variable.
Associations between the screening performance of each individual condition (yes/no), including FGM, and patients' age (in years) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for one of the seven infections and/or screened for female genital mutilation/no-if the patient was not tested) as the outcome variable and patients' age as the predictor variable.
Associations between the screening performance of each individual condition (yes/no), including FGM, and the time that patients have been registered in the Spanish Health System (in years) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for one of the seven infections and/or screened for female genital mutilation/no-if the patient was not tested) as the outcome variable and time registered in the Spanish Health System as the predictor variable.
Associations between the screening performance of each individual condition (yes/no), including FGM, and patients' sex (female/male) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes- yes-if the patient has been tested for one of the seven infections and/or screened for female genital mutilation/no-if the patient was not tested) as the outcome variable and patients' sex as the predictor variable.
Associations between the screening performance of each individual condition (yes/no), including FGM, and patients' area of birth (Africa/Latin America/Asia/Eastern Europe) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for one of the seven infections and/or screened for female genital mutilation/no-if the patient was not tested) as the outcome variable and patients' area of birth as the predictor variable. The areas of birth will be based in the geographical division of the United Nations Statistical Division.
Associations between the screening performance of each individual condition (yes/no), including FGM, and the region where the PCC is located (Terres de l'Ebre/Lleida/Tarragona/Costa de Ponent) will be analysed using data collected in the SISAP database | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for one of the seven infections and/or screened for female genital mutilation/no-if the patient was not tested) as the outcome variable and the region of the PCC as the predictor variable.
Associations between the screening performance of each individual condition (yes/no), including FGM, and the type of region where the PCC is located in Catalonia, Spain (urban/rural) will be analysed using the data collected in the SISAP database | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for one of the seven infections and/or screened for female genital mutilation/no-if the patient was not tested) as the outcome variable and the type of region of the PCC as the predictor variable.
Associations between the screening performance each individual condition (yes/no), including FGM, and if the patient fulfilled the criteria of the screening recommendation (yes/no) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for one of the seven infections and/or screened for female genital mutilation/no-if the patient was not tested) as the outcome variable and fulfilled the criteria of the screening recommendation (yes- if the patient had the criteria of being tested for at least one infection, criteria generated by the algorithm of the ISMiHealth software using the variables country of birth, age and sex/no- if the patient did not meet the criteria) as the predictor variable.
Associations between the screening performance of each individual condition (yes/no), including FGM, and the arm of the study (Intervention/Control) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for one of the seven infections and/or screened for female genital mutilation/no-if the patient was not tested) as the outcome variable and the arm of the study as the predictor variable.
Associations between the screening performance of each individual condition (yes/no), including FGM, and patients' immunosuppression status (yes/no) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for one of the seven infections and/or screened for female genital mutilation/no-if the patient was not tested) as the outcome variable and patients' immunosuppression status (yes- if the patient has an ICD-code diagnosis of an immunosuppressive disorder and/or have a prescription of an immunosuppressive drug/no- if the patient is not immunosuppressed) as the predictor variable.
Associations between the screening performance of each individual condition (yes/no), including FGM, and the presence of another condition (yes/no) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for one of the seven infections and/or screened for female genital mutilation/no-if the patient was not tested) as the outcome variable and the presence of another condition (yes- if the patient has an ICD-code of another condition [co-morbidity]/no- if the patient does not present another condition) as the predictor variable.
Associations between the screening performance of HIV (yes/no) and the CD4 cell count (cell/µL) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for HIV during the study period/no-if the patient was not tested) as the outcome variable and the CD4 cell count as the predictor variable.
Associations between the screening performance of HIV (yes/no) and the viral load (copies/mL) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for HIV /no-if the patient was not tested) as the outcome variable and the viral load as the predictor variable.
Associations between the screening performance of HBV and/or HCV (yes/no) and the levels of platelets (U/µL) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for HBV and/or HCV /no-if the patient was not tested) as the outcome variable and the levels of platelets as the predictor variable.
Associations between the screening performance of HBV and/or HCV (yes/no) and the levels of transaminases (U/L) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for HBV and/or HCV /no-if the patient was not tested) as the outcome variable and the levels of transaminases as the predictor variable.
Associations between the screening performance of HBV and/or HCV (yes/no) and the levels of bilirubin (mg/dL) will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for HBV and/or HCV /no-if the patient was not tested) as the outcome variable and the levels of bilirubin as the predictor variable.
Associations between the screening performance of HBV and/or HCV (yes/no) and the levels of clotting parameters [such as prothrombin (seconds), fibrinogen (mg/dL), among others] will be analysed using the data collected from the EPR system | Through study completion, 1 year.
  Bivariate and multivariate analysis (Fisher's exact tests, Chi-square tests and/or logistic regressions) will be performed using the screening performance of each individual condition (yes-if the patient has been tested for HBV and/or HCV /no-if the patient was not tested) as the outcome variable and the levels of clotting parameters as the predictor variable.
Number of diagnosed individuals with follow-up visits in the hospital of reference | Through study completion, 1 year.
  The number of migrant patients under follow-up in the hospital after a diagnosis of an infection or FGM will be estimated using the Minimum basic dataset (MBDS).
Number of diagnosed individuals under treatment | Through study completion, 1 year.
  The number of migrant patients under treatment after a diagnosis will be estimated using data from the EPR systems and the MBDS.

OTHER OUTCOMES:
Prevalence of each individual condition in the migrant population | Through study completion, 1 year.
  The prevalence of each condition will be estimated using as the denominator the total number of tested migrant patients for that specific condition. Then, these results will be compared with other studies and country registries.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Requena Méndez, PhD, Principal Investigator — Barcelona Institute for Global Health
Locations (2):
- Spain (2):
  - Servicio Andaluz de Salud (SAS) (administration of the participant PCCs in Andalusia), Almería, Andalusia
  - Institut Català de la Salut (ICS) (administration of the participant PCCs in Catalonia), Tortosa, Catalonia

IPD SHARING:
Plan to Share IPD: Yes
The project involves handling personal data that are routinely collected in healthcare services. Data will be obtained retrospectively and study variables will be pseudo-anonymized by the IT staff of each healthcare system. Pseudo-anonymized data will be stored and secured in the local server of ISGlobal (VPN) and only participating investigators will have access to it. An adequate documentation of (meta) data will facilitate identification and support effective reuse of research data. A standardized communications protocol to retrieve (meta) data will be generated.
  Anonymous data will be stored in a repository in ISGlobal's data centre (Carrer Dr. Aiguader, 88) for 10 years. Only encrypted data will be transferred to third parties and other countries, solely for the same purpose of the study described and would guarantee confidentiality.
  Data will be findable for the research community through the trial registration and scientific publications.
Supporting Information: Study Protocol, SAP
Time Frame: Data and metadata will be deposited into ISGlobal's repository at the time of publication or by the end of the project period, whichever comes first. After 10 years, all data will be eliminated and destroyed.
Access Criteria: Pseudo-anonymized data in ISGlobal's VPN will only be accessed by investigators. In addition, a password will be requested to all researchers in order to access the data, registering any access.
  Anonymous data will be available from the corresponding author upon reasonable request.

REFERENCES:
- [Background] Sequeira-Aymar E, diLollo X, Osorio-Lopez Y, Goncalves AQ, Subira C, Requena-Mendez A. [Recommendations for the screening for infectious diseases, mental health, and female genital mutilation in immigrant patients seen in Primary Care]. Aten Primaria. 2020 Mar;52(3):193-205. doi: 10.1016/j.aprim.2019.02.005. Epub 2019 Apr 25. Spanish. PMID 31029458
- [Background] Sequeira-Aymar E, Cruz A, Serra-Burriel M, di Lollo X, Goncalves AQ, Camps-Vila L, Monclus-Gonzalez MM, Revuelta-Munoz EM, Busquet-Sole N, Sarriegui-Dominguez S, Casellas A, Llorca MRD, Aguilar-Martin C, Jacques-Avino C, Hargreaves S, Requena-Mendez A; CRIBMI (IS-MiHealth) Working Group. Improving the detection of infectious diseases in at-risk migrants with an innovative integrated multi-infection screening digital decision support tool (IS-MiHealth) in primary care: a pilot cluster-randomized-controlled trial. J Travel Med. 2022 Nov 4;29(7):taab100. doi: 10.1093/jtm/taab100. PMID 34230959
- [Derived] Cruz A, Cuxart-Graell A, Goncalves AQ, Vazquez-Villegas J, Vallejo-Godoy S, Salas-Coronas J, Piqueras N, Martinez-Torres S, Artigues-Barbera E, Rando-Matos Y, Margalejo AA, Vizcaino J, Requena P, Martinez-Perez A, Ferrer E, Mendez-Boo L, Coma E, Luzon-Garcia MP, Sequeira-Aymar E, Casellas A, Vazquez M, Jacques-Avino C, Medina-Perucha L, Sicuri E, Evangelidou S, Aguilar Martin C, Requena-Mendez A. Delivering an innovative multi-infection and female genital mutilation screening to high-risk migrant populations (ISMiHealth): study protocol of a cluster randomised controlled trial with embedded process evaluation. BMJ Open. 2024 Nov 4;14(11):e078337. doi: 10.1136/bmjopen-2023-078337. PMID 39496367

DOCUMENTS (2):
  • Study Protocol (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT05868005/Prot_003.pdf
  • Statistical Analysis Plan (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/05/NCT05868005/SAP_002.pdf